CLINICAL TRIAL: NCT03699579
Title: Patients Characteristics, Treatment Utilization, Costs and Outcomes in Patients With Advanced or Metastatic Renal Cell Carcinoma (RCC) Who Received at Least One Prior Vascular Endothelial Growth Factor (VEGF)-Targeted Therapy in Taiwan
Brief Title: Pharmaco-Economic Study of Treatment Options in Patients With Advanced RCC
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-TW-60000-022
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Renal Cell Carcinoma Metastatic; Renal Cell Carcinoma
Keywords: advanced or metastatic renal cell carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a retrospective cohort study aiming to collect data on patients' characteristics, resource utilization, adverse events management and calculate costs attributed to current treatments of advance RCC patients who have received at least one prior VEGF-targeted therapy in Taiwan from National Health Insurance (NHI) perspective.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of clear-cell renal cell carcinoma
* Patients with evidence of metastatic disease
* Patients who have received at least one previous VEGFR-targeted therapy, i.e sunitinib, pazopanib or sorafenib
* Patients who received care at the selected medical centers, utilizing the National Health Insurance (NHI) reimbursed system at the time of the disease

Exclusion Criteria:

* Patients enrolled in any clinical trial involving anti-cancer therapy
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital chart review study
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2019-06-23 (Actual)

PRIMARY OUTCOMES:
Medication usage | From start point for 2.5 months
Treatment's duration | From start point for 2.5 months

SECONDARY OUTCOMES:
Cost of medication used | From start point for 2.5 months
Costs of adverse event management | From start point for 2.5 months
  (total calculated costs attributed to Adverse Effects (AEs) management according to the attached list of adverse events
Frequency of health resource usage | From start point for 2.5 months
  Outpatient department visits, CT scan, blood test number and types
Cost of health resource usage | From start point for 2.5 months
  Outpatient department visits, CT scan, blood test number and types

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei